CLINICAL TRIAL: NCT03960398
Title: Incidence of Iatrogenic Diseases on Toulon-La Seyne Sur Mer Hospital Emergency Consultations During Summer 2018
Brief Title: Incidence of Iatrogenic Diseases on Hospital's Emergency Consultations
Acronym: EIU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-CHITS-02
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Iatrogenic Disease
Keywords: iatrogenic; emergency; incidence; adverse drug reaction
MeSH Terms: conditions — Iatrogenic Disease; Emergencies; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients concerned by iatrogenic diseases: Patients living in the South-East of France and consulting in the emergency department of Toulon La Seyne sur Mer hospital for iatrogenic diseases
  Interventions: Drug: Iatrogenic disease impact on emergency consultations

INTERVENTIONS:
Drug: Iatrogenic disease impact on emergency consultations — Determination of the proportion of emergency consultations linked to iatrogenic diseases

SUMMARY:
French population grows older year after year: 24.3% people were over 60 years old in 2006 against 20.6% in 2000 and the expected number might be over 33% in 2050.

The elderly suffer from lots of illnesses, so they usually take lots of drugs. Therefore, this drug use is most likely to have adverse drug reactions.

Finally, according to Health Ministry, the number of emergency department consultations doubled from 1996 to 2016.

Consequently, it is interesting to study the impact of drug iatrogenic effects on emergency consultations.

It would help to prevent these adverse drug reactions as we prescribe those drugs : First, do not harm.

DETAILED DESCRIPTION:
This will be a retrospective study.

The number of patients will be defined by the number of visits during a random draw of 10 emergency department consultation days between 21st June 2018 and 22nd September 2018 in Toulon - La Seyne sur Mer public hospital.

There are between 100 and 300 emergency department consultations per day in this hospital so the estimated number of patients will be between 1000 and 3000.

Every patient who came to hospital for a consultation in emergency department during this period of time will be included in the study except those who expressed their opposition to their data collection and treatment.

Each patient will be anonymized with a code defined as follows : N(ame) L(ast name) 001 (chronological inclusion number)

Information of the patients involved in adverse drug reactions will be extracted and a description of this patient sample will be made.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years old
* Consultation in emergency department of Sainte Musse or La Seyne-sur-Mer hospital between 21st june 2018 and 22nd september 2018 included
* Consultation of the patient in emergency department during the 10 day random draw of the research (from 00h01 to 23h59)
* Consultation in emergency department because of a iatrogenic reason

Exclusion Criteria:

* Dead patients
* Patient's opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adults living in the south-east of France and consulting the emergency department of Toulon - La Seyne sur Mer public hospital
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients coming to emergency department because of an adverse drug reaction | 10 days (chosen at random between 21st June and 22nd September 2018)
  We will study each case and determine whether the consultation in the emergency department is due to adverse drug reaction or not.Number of patients having an emergency department consultation because of an adverse drug reaction divided by the total number of patients having an emergency department consultation during the same period of time.

SECONDARY OUTCOMES:
Average of patient age among the patients consulting because of an adverse drug reaction | 10 days
  Average and standard deviation of patient age among the patients consulting in emergency department because of an adverse drug reaction.
Proportion of male and female patients consulting because of an adverse drug reaction | 10 days
  Number of male and female patients consulting in emergency department because of an adverse drug reaction divided by the total number of patients consulting in emergency department because of an adverse drug reaction.
Number of treatments administered to patients who consult because of an adverse drug reaction | 1 day
  Number of treatments patients were taking when they arrived in emergency department for a consultation because of an adverse drug reaction
Frequency of the drugs leading to a consultation in emergency department because of an adverse drug reaction | 10 days
  For each drug leading, during the 10 chosen days, to a consultation because of an adverse reaction, number of times when this drug was at the origin of a consultation

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana PLATINO, MD, Study Director — Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal de Toulon - La Seyne sur Mer, La Seyne-sur-Mer, Var
  - Centre Hospitalier Intercommunal de Toulon - La Seyne sur Mer, Toulon, Var

IPD SHARING:
Plan to Share IPD: No